CLINICAL TRIAL: NCT06119594
Title: Contribution of the Evaluation of Body Composition by Connected Scale in the Effectiveness of a Reconditioning Program Through Physical Activity Adapted for Patients Suffering From Chronic Diseases
Acronym: COCORAPA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hôpital Lariboisière Fernand Widal (Other); Hotel Dieu Hospital (Other); Withings (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP230549; 2023-A01156-39 (Other: IDRCB)
Record Dates: First submitted 2023-10-16; First posted 2023-11-07 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Disease
Keywords: physical activity rehabilitation program; Connected scale
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Comparative, controlled, randomized by cluster 1:1 open, in two parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard follow-up group (No Intervention): Routine care
- Connected scale group (Experimental): Routine care + use of connected scale during 6 months
  Interventions: Device: Body Comp Pro connected scale (Withings manufacturer)

INTERVENTIONS:
Device: Body Comp Pro connected scale (Withings manufacturer) — Patients in the intervention group will use the connected scale at a minimum frequency of once a week from receipt of the scale and throughout their participation in the research (6 months)
  Arms: Connected scale group

SUMMARY:
The goal of this interventional study is to evaluate the impact of the use of a connected impedance scale on the physical and mental quality of life of patients suffering from chronic diseases and participating in a physical activity rehabilitation program. The main objective is to know if a regular monitoring of the evolution of body composition parameters recorded by the connected scale would allow patients participating in the Physical Activity rehabilitation program at Hôtel-Dieu to follow in real time the effects of such program, not on weight itself but on body composition, and that this would contribute to a better perception of physical and mental quality of life at the end of the program 90 Participants will be randomized in two groups :

* Control group (N = 45) : routine care
* Interventionnal group (N=45) : routine care + use of connected scale All participants will undergo physical activity rehabilitation program during 6 weeks.

Patients will be see again at 6 months, and the following parameters will be comparer between the two groups :

* SF-36 questionnaire
* Ricci & Gagnon questionnaire
* 6MWT
* 30 sec sit-to stand test
* Ito-Shirado test
* Sorensen test
* Handgrip test
* MaxV02

ELIGIBILITY:
Inclusion Criteria:

* Patient (male or female) aged 18 and over
* Patient able to express free, informed and written consent
* Patient participating in the physical activity rehabilitation program at the CIMS of the Hôtel Dieu
* Patient suffering from a known, stable and diagnosed chronic disease
* Patient autonomous in taking treatments for their ALD
* Patient affiliated to a social security system

Exclusion Criteria:

* Patient under legal protection (guardianship, curatorship)
* Patient deprived of liberty by a judicial or administrative decision
* Patient with functional limitations that do not allow a physical assessment or result in a walking distance < 350 m during the HDJ for admission to the program
* Patient with suspected cardiac pathology during the HDJ for admission to the program
* Patient with episode of decompensation or exacerbation
* Patient with a pacemaker or implantable automatic defibrillator
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the physical and mental quality of life score using the Short Form 36 questionnaire at 6 months for each patient. | 6 months from initiation of physical activity rehabilitation program
  Short Form 36 questionnaire (0 - 100 ; Higher mean better outcome)

SECONDARY OUTCOMES:
Measurement of the physical and mental quality of life score using the Short Form 36 questionnaire at 6 weeks for each patient. | 6 weeks from initiation of physical activity rehabilitation program
  Short Form 36 questionnaire (0 - 100 ; Higher mean better outcome)
Measurement of daily physical activity level by the Ricci & Gagnon questionnaire at 6 months for each patient | 6 months from initiation of physical activity rehabilitation program
  Ricci & Gagnon questionnaire (9 - 45 ; Higher mean better outcome)
Measurement of 6 minute walk test (6MWT) at 6 months for each patient | 6 months from initiation of physical activity rehabilitation program
  6 minute walk test (Higher mean better outcome)
Measurement of 30 sec sit-to-stand test at 6 months for each patient | 6 months from initiation of physical activity rehabilitation program
  30 sec sit-to-stand test (Higher mean better outcome)
Measurement of Ito-Shirado test at 6 months for each patient | 6 months from initiation of physical activity rehabilitation program
  Ito-Shirado test (Higher mean better outcome)
Measurement of Sorensen test at 6 months for each patient | 6 months from initiation of physical activity rehabilitation program
  Sorensen test (Higher mean better outcome)
Measurement of Handgrip test at 6 months for each patient | 6 months from initiation of physical activity rehabilitation program
  Handgrip test (Higher mean better outcome)
Measurement of VO2max at 6 months for each patient | 6 months from initiation of physical activity rehabilitation program
  VO2

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigations en Médecine du Sport - Hôpital Hôtel Dieu, Paris, France

IPD SHARING:
Plan to Share IPD: No